CLINICAL TRIAL: NCT04085341
Title: A Phase 2a Multicenter Study Evaluating the Safety, Tolerability, and Pharmacodynamics of Sunitinib Malate Depot Formulation (GB-102) in Subjects With Diabetic Macular Edema (DME) and Retinal Vein Occlusion (RVO)
Brief Title: A Depot Formulation of Sunitinib Malate (GB-102) in Subjects With Diabetic Macular Edema and Retinal Vein Occlusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Graybug Vision (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBV-102-003
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Macular Edema; Retina Vein Occlusion
Keywords: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Sunitinib

STUDY DESIGN:
Intervention Model Description: Parallel-arm design
Masking Description: Open-label study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GB-102 Dose 1 (1 mg) (Experimental): Participants will receive intravitreal (IVT) GB-102 (1 mg) in the study eye at Baseline.
  Interventions: Drug: GB-102
- GB-102 Dose 2 (2 mg) (Experimental): Participants will receive intravitreal (IVT) GB-102 (2 mg) in the study eye at Baseline.
  Interventions: Drug: GB-102

INTERVENTIONS:
Drug: GB-102 — Intravitreal injection of GB-102
  Other Names: Sunitinib malate

SUMMARY:
Phase 2a multicenter, open-label, parallel-arm design study to evaluate the safety, tolerability and pharmacodynamics of a single intravitreal injection comparing 2 dose levels of GB-102 on subjects with Diabetic Macular Edema and Retinal Vein Occlusion

DETAILED DESCRIPTION:
Phase 2a multicenter, open-label, parallel-arm design study to evaluate the safety, tolerability and pharmacodynamics of a single intravitreal injection comparing 2 dose levels (1 mg and 2 mg) of GB-102 on subjects with Diabetic Macular Edema and Retinal Vein Occlusion who have received prior treatment with anti-vascular endothelial growth factor (VEGF)

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 21 years of age
* Known diagnosis of macular edema secondary to diabetic macular edema or retinal vein occlusion treated with at least 3 prior IVT injections of an anti-VEGF agent (aflibercept, bevacizumab, or ranibizumab)
* Demonstrated response to prior anti-VEGF treatment since diagnosis
* BCVA of 31 letters or better

Exclusion Criteria:

* History, within 6 months prior to screening, of any of the following: myocardial infarction, any cardiac event requiring hospitalization, treatment for acute congestive heart failure, transient ischemic attack, or stroke
* Uncontrolled hypertension, diabetes mellitus or IOP
* Chronic renal disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Graybug Vision, Inc.
Locations (6):
- United States (6):
  - Retinal Research Institute, Phoenix, Arizona
  - Southern Retina, Savannah, Georgia
  - Eye Care Institute, Louisville, Kentucky
  - Boston Retina, Boston, Massachusetts
  - Sierra Eye Associates, Reno, Nevada
  - Texoma Retina Center, Denison, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GB-102 Dose 1 (1 mg) | GB-102 Dose 2 (2 mg)
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GB-102 Dose 1 (1 mg) | GB-102 Dose 2 (2 mg) | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (13.83) | 65.1 (10.5) | 64.9 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 11 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Adverse Events (AEs) Across All Study Visits
Description: Number of subjects with an adverse event across all study visits
Time Frame: Baseline through Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | GB-102 Dose 1 (1 mg) | GB-102 Dose 2 (2 mg)
Number analyzed (Participants) | 10 | 11
Participants | 7 | 10

2. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) (ETDRS) at All Study Visits
Description: BCVA = best corrected visual acuity; ETDRS = early treatment of diabetic retinopathy
  BCVA = 0 (worst) to 100 (best)
  Assessment of change in BCVA (ETDRS letter score) from baseline at all visits
Time Frame: Baseline to Month 6
Measure: Mean (Full Range); unit: letters
Arm/Group | GB-102 Dose 1 (1 mg) | GB-102 Dose 2 (2 mg)
Number analyzed (Participants) | 10 | 11
letters | -10.4 [-32 to 4] | -16.7 [-75 to 15]

3. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness (CST) (SD-OCT) at All Study Visits
Description: CST = central subfield thickness
  SD-OCT = spectral domain-optical coherence tomography
  Assessment of change in CST (μm) measurement from baseline at all visits
Time Frame: Baseline to Month 6
Measure: Mean (Full Range); unit: micrometers
Arm/Group | GB-102 Dose 1 (1 mg) | GB-102 Dose 2 (2 mg)
Number analyzed (Participants) | 10 | 10
micrometers | 131.0 [-13.0 to 374.0] | -37.4 [-198.0 to 73.0]

4. Secondary Outcome: Time to Rescue Treatment
Description: Assessment of time to rescue treatment over 6 months of treatment
Time Frame: Baseline through Month 6
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | GB-102 Dose 1 (1 mg) | GB-102 Dose 2 (2 mg)
Number analyzed (Participants) | 10 | 11
days | 90 [60 to 120] | 120 [60 to NA] — NA = not applicable/ not estimable due to small sample size and insufficient number of participants who needed rescue treatment.

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from baseline for the duration of a subject's participation in the study (up to 180 days). AEs are reported as treatment-emergent.
Description: An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug-related. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. Ocular AEs are presented for both study eye and non-study eye combined.
Arm/Group | GB-102 Dose 1 (1 mg) | GB-102 Dose 2 (2 mg)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/10 | 2/11
Other Adverse Events (participants affected / at risk) | 7/10 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GB-102 Dose 1 (1 mg) (N=10) | GB-102 Dose 2 (2 mg) (N=11)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Corneal Oedema (Eye disorders) | 0 (0) | 1 (1)
Visual Impairment (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GB-102 Dose 1 (1 mg) (N=10) | GB-102 Dose 2 (2 mg) (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Vascular Malformation Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood Potassium Decreased (Investigations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (2) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Posterior Capsule Opacification (Eye disorders) | 0 (0) | 1 (2)
Retinal Aneurysm (Eye disorders) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 2 (2) | 3 (3)
Visual Acuity Reduced (Eye disorders) | 2 (2) | 3 (3)
Vitreous Floaters (Eye disorders) | 2 (2) | 3 (3)
Macular Edema (Eye disorders) | 4 (4) | 0 (0)
Vision Blurred (Eye disorders) | 2 (2) | 1 (1)
Visual Impairment (Eye disorders) | 1 (1) | 1 (2)
Iridocyclitis (Eye disorders) | 0 (0) | 2 (2)
Swelling of Eyelid (Eye disorders) | 1 (1) | 1 (1)
Cataract Nuclear (Eye disorders) | 0 (0) | 1 (1)
Conjunctival Irritation (Eye disorders) | 0 (0) | 1 (1)
Corneal Edema (Eye disorders) | 0 (0) | 1 (1)
Eye Irritation (Eye disorders) | 0 (0) | 1 (1)
Eye Edema (Eye disorders) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 0 (0) | 1 (1)
Lacrimation Increased (Eye disorders) | 0 (0) | 1 (1)
Ocular Hyperaemia (Eye disorders) | 1 (2) | 0 (0)
Pterygium (Eye disorders) | 1 (1) | 0 (0)
Punctate Keratitis (Eye disorders) | 1 (1) | 0 (0)
Pupils Unequal (Eye disorders) | 0 (0) | 1 (1)
Product Residue Present (Investigations) | 2 (2) | 6 (8)
Intraocular Pressure Increased (Investigations) | 0 (0) | 2 (4)
Vital Dye Staining Cornea Present (Investigations) | 0 (0) | 1 (1)
Chorioretinitis (Infections and infestations) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Too few subject numbers divided across multiple indications. The trial was conducted in 21 subjects with Diabetic Macular Edema, Branch Retinal Vein Occlusion and Central Retinal Vein Occlusion divided between two doses. Subjects had variable disease control and duration prior to entry.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any investigator wishing to publish or present any study finding must present a manuscript or abstract to Graybug Vision 120 days prior to submission for publication or presentation to provide Graybug Vision an opportunity for review and comment.

DOCUMENTS (2):
  • Study Protocol (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT04085341/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT04085341/SAP_001.pdf